CLINICAL TRIAL: NCT06318338
Title: Virtual Reality to Promote Mindfulness and Relaxation Prior to Radiation Simulation: a Prospective Pilot Feasibility Study
Brief Title: Virtual Reality to Promote Relaxation Prior to Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Michael LaRiviere, MD, Assistant Professor of Radiation Oncology, Abramson Cancer Center at Penn Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCC 14523; 854756 (Other: Penn IRB)
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: Virtual Reality; Relaxation; Mindfulness
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Reality Program (Experimental): This is a single arm study. All participants will participate in the study intervention, which involves experiencing a virtual reality program.
  Interventions: Other: Virtual Reality Program

INTERVENTIONS:
Other: Virtual Reality Program — Study participants will be provided a HTC or Pico VR head-mounted device (HTC Flow, HTC Focus or Pico Neo Pro) which will be fitted for comfort. Patients will remain seated for the entirety of the VR program. The program generally takes about ten minutes to complete but may last up to 11 minutes. The program displays a relaxing environmental setting with narration based in mindfulness meditation principles. Subjects will be prompted to practice breathing exercises designed to relax and reduce anxiety.

SUMMARY:
The purpose of this study is to assess the feasibility of a pre-simulation virtual reality (VR) platform designed to promote relaxation for cancer patients planned for radiation therapy (RT).

DETAILED DESCRIPTION:
The purpose of this prospective feasibility study is to assess the implementation of a VR-based intervention in patients who are pending initiation of RT. The investigators hypothesize that this intervention will be safe and feasible. If 75% of enrolled patients complete the VR intervention (defined as at least 8 min before permanent discontinuation), then feasibility will be met. Ten minutes' length is likely to be tolerated by most patients and likely to provide benefit. The maximum length of the VR video is 11 minutes. Patients will still be evaluable after 8 minutes of the video as this provides ample time to practice mindfulness based breathing exercises.

As this is a feasibility study, investigators and participants will not be blinded to study procedures. Potential study participants will be adult patients who are undergoing simulation for radiation treatment planning at the Perelman Center for Advanced Medicine at Penn Medicine. This is a single site study. No interim analyses or sub-studies are planned. Based on the expected accrual of 25 patients, futility and early termination will be triggered if 6 participants fail to meet the conditions described above.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand, read or speak English sufficient for signing of informed consent and completion of study assessments
2. Patients scheduled for simulation for radiation treatment planning at Perelman Center for Advanced Medicine (PCAM)
3. Adults, at least 18 years of age
4. Performance Status (ECOG) 0-2

Exclusion Criteria:

1. Prior radiotherapy
2. History of motion sickness, car sickness, vertigo, migraines, or light sensitivity within the last 6 months
3. History of epilepsy and seizures
4. Current nausea, vomiting, dizziness, lightheadedness, monocular vision or hearing loss that is not treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of a pre-simulation VR platform prior to radiation | 12 months
  Feasibility based on the ability of at least 75% patient VR completion rate. Based on the expected accrual of 25 patients, futility and early termination will be triggered if six participants fail to meet the conditions described above.

SECONDARY OUTCOMES:
Patient feedback on pre-simulation VR program | 12 months
  To collect patient feedback on the usability of and overall satisfaction with the VR program prior to simulation. Post-intervention survey designed to collect qualitative and quantitative patient feedback.
Patient situational anxiety prior to and after use of VR program (HADS) | 12 months
  To evaluate patient-reported situational anxiety levels prior to and after use of the VR headset.
  Measure baseline score on Hospital Anxiety and Depression Scale (HADS). The HADS is a 14-item scale with seven items for each anxiety and depression. Subscale scores greater than 8 denotes anxiety or depression.
Patient situational anxiety prior to and after use of VR program (STAI-6) | 12 months
  To evaluate patient-reported situational anxiety levels prior to and after use of the VR headset.
  Measure change in the State-Trait Anxiety Inventory (STAI-6) score at baseline and after VR intervention. The STAI-6 is adapted from the original 20-item STAI. The original STAI scores range from 20-80. A score of 40 or higher is correlated with high anxiety. The STAI-6 consists of six questions rated on a 1-4 Likert scale creating a score range from 6 to 24. In order to generate scores compatible with the original STAI, STAI-6 scores will be multiplied by 20 and divided by 6 to give a range between 20-80.

CONTACTS AND LOCATIONS:
Overall Officials: Michael LaRiviere, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No